CLINICAL TRIAL: NCT05016752
Title: Application of Nanopore Sequencing in Newly Diagnosed Acute Myeloid Leukemia Patients With Neutropenia and Bloodstream Infection: a Prospective Multicenter Observational Clinical Study
Brief Title: Application of Nanopore Sequencing in Newly Diagnosed Acute Myeloid Leukemia Patients With Bloodstream Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021174
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Blood Stream Infection; Gut Microbiota; Acute Myeloid Leukemia
Keywords: Nanopore sequencing; Blood culture
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, faeces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute myeloid leukemia (AML) patients are prone to blood stream infection (BSI) due to bone marrow suppression, oral and gastrointestinal mucositis, endovascular tubes, and the application of a large number of broad-spectrum antibiotics. The associated mortality rate is as high as 7.1 %-42%. The use of antibiotics within one hour after the first observation of hypotensive symptoms can guarantee a 79.9% survival rate. For every hour of delay, the patient's survival rate will drop by 7.6%. At present, the blood culture test cycle is long and the positive rate is low. Other infection-related indicators (PCT, CRP) or next-generation sequencing are not highly specific and easy to be misdiagnosed. X-ray, CT and other examinations only have a certain auxiliary value for the infected site. We need new diagnostic tools to accurately identify pathogens. Nano-seq is a next-generation sequencing technology for single-molecule, real-time sequencing and analysis. With ultra-long sequencing read length, it can quickly and accurately identify BSI pathogens types, and give appropriate drug sensitivity results based on drug resistance genes to meet the needs of 99.9% pathogen screening. At the same time, we hope to conduct a prospective evaluation to target high-risk groups of AML prone to BSI in the early stage. The intestine is the body's largest immune organ and the largest reservoir of microbial pathogens. The expansion of certain gut microbiota usually precedes BSI. If there is a correlation between the gut microbiota and MDR-BSI, the colonization and changes of the intestinal flora can be used to predict the risk of BSI in patients during treatment, and preventive measures such as early decolonization or biological intervention will reduce the risk of infection in the future. Combined with Nano-seq and various existing clinical pathogen detection technologies to reduce the occurrence and progress of clinical BSI.

DETAILED DESCRIPTION:
For AML patients with bloodstream infections, we analyzed and compared the sensitivity, specificity, and consistency of Nano-seq and traditional blood culture tests, and evaluated the advantages of Nano-seq for clinical diagnosis and treatment guidance of newly-treated AML bloodstream infections. At the same time, the homology analysis of gut microbiota and bloodstream infection strains was carried out to explore the correlation between gut microbiota and bloodstream infection in newly treated AML patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML according to the WHO (2016) classification of acute myeloid leukemia.
* No history of previous chemotherapy or target therapy.
* Neutrophil deficiency (ANC<0.5x10^9/L) with the first time fever(Oral temperature >=38.3 degree C or axillary temperature >=38.0 degree C) accompanied by chills or hemodynamic instability(BP <=90/60mmHg）
* Ability to comprehend the investigational nature of the study and provide informed consent.

Exclusion Criteria:

* Patients have a history of chemotherapy or target therapy.
* Patients with other commodities that the investigators considered not suitable for the enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed acute myeloid leukemia patients with neutropenia and bloodstream infection
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Nano-seq group compared to blood culture group | Within 2 week of sampling.
  Proportion of samples where Nano-seq detects a pathogenic micro-organism that has been identified by blood culture diagnostic pathway.
Specificity of Nano-seq group compared to blood culture group | Within 2 week of sampling.
  Proportion of samples where Nano-seq does not detect a micro-organism where blood culture diagnostic pathway has also not detected a micro-organism.
Level of agreement between Nano-seq group and blood culture group | Within 2 week of sampling.
  Proportion of samples where the two methods produce the same result.

SECONDARY OUTCOMES:
To compare the detection time, the intensity, duration and cost of antibiotics,length and cost of hospitalization between the Nano-seq group and blood culture group | 3 months
  To assess the difference between Nano-seq group and blood culture group in terms of timeliness and hospitalization costs
Analyze the homology of the gut microbiota of patients with bloodstream infections and the detected strains | 3 months
  To assess the source of bloodstream infection and record the clinical high-risk factors and treatment outcomes
Intestinal flora OTU clustering, genus abundance, Alpha diversity, Beta diversity, differences between LEfse groups, baseline value and subsequent changes in the prediction of the metabolic function of the gut microbiota | 3 months
  To assess the correlation between colonization and changes of gut microbiota and bloodstream infections

CONTACTS AND LOCATIONS:
Overall Officials: Haiping Dai, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China